CLINICAL TRIAL: NCT02875093
Title: Phase 1 Study of ADI-PEG 20 Plus Low Dose Cytarabine in Older Patients With Acute Myeloid Leukemia
Brief Title: Ph 1 Study of ADI-PEG 20 Plus Low Dose Cytarabine in Older Patients With AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Termination
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2016-001
Record Dates: First submitted 2016-08-09; First posted 2016-08-23 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ADI PEG20; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADI-PEG 20 Plus Low Dose Cytarabine (Other): This is a phase 1, open label trial of ADI-PEG 20 (18 and 36 mg/m2) weekly in combination with low-dose cytarabine (20 mg BID [twice daily] for 10 days, every 28 days)
  Interventions: Drug: ADI-PEG 20; Drug: Cytarabine

INTERVENTIONS:
Drug: ADI-PEG 20 — Investigational Medicine
Drug: Cytarabine — low-dose cytarabine 20 mg BID twice daily for 10 days, every 28 days

SUMMARY:
Assessment of safety and tolerability of drug combination and determine time on treatment, Overall survival (OS) and response rate with patient disease burden, and type of disease

ELIGIBILITY:
Inclusion Criteria:

1. AML diagnosed by morphologic (with >20% blasts in blood or bone marrow) and histochemical and/or cell surface marker criteria.
2. Patients with AML must fall into one of the following:

   1. Patients with AML (i.e., > 20% bone marrow blasts) who are deemed unfit* for intensive chemotherapy with refractory or relapsed disease. The patients must have been refractory to at least one cycle of cytarabine containing regimens or at least two cycles of azacitidine or similar hypomethylating agents.
   2. Patients with untreated AML (i.e., > 20% bone marrow blasts) with intermediate risk karyotype (MRC risk group) who are deemed unfit for intensive chemotherapy.
   3. Patients with untreated AML with adverse risk karyotype (MRC risk group) who are deemed unfit for intensive chemotherapy and who are intolerant of azacitidine (or other hypomethylating agents) or who are unable to access azacitidine or other hypomethylating agents.

      * Patients unfit for conventional intensive chemotherapy are defined as having at least one of the following based on the conceptual criteria of Ferrara (2013):

        1. Advanced age (over 75 years).
        2. Cardiac impairment with ejection fraction ≤ 50% or heart failure (NYHA class 2) or ischemic heart disease with stable angina.
        3. Pulmonary impairment: chronic obstructive pulmonary disease (COPD) stage 1-2 (forced expiratory volume in one second [FEV1] > 49%) or other comparable respiratory disease with forced vital capacity (FVC) > 50%.
        4. Hepatic comorbidity with Child-Pugh grade A cirrhosis
        5. Chronic kidney disease stage 3 but with creatinine clearance > 30 mls/min
        6. Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy.
3. Age > 17 years.
4. ECOG performance status of 0-2.
5. Bone marrow aspirate and/or biopsy for testing for ASS1-deficiency. This must be a fresh sample obtained after any prior chemotherapy and before enrollment in this study. ASS1-deficiency is not required for study entry, but the fresh bone marrow sample must be processed either before or within 1 week of first study dose (see Section 10 for more details).

Exclusion Criteria:

A subject will not be eligible for study participation if he/she meets any of the exclusion criteria:

1. Patients with uncontrolled infections requiring intravenous (IV) antibiotic/antiviral therapy are not eligible for entry onto the study; patients on prophylactic antibiotics or antivirals are acceptable.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina, ventricular cardiac arrhythmia (other than ventricular ectopy), severe pulmonary comorbidity: COPD grade 3-4 (FEV1 <50%) or other comparable documented pulmonary disease with FVC <50%, or dyspnea at rest or requiring oxygen at home, cognitive impairment: current mental illness requiring psychiatric hospitalization, institutionalization or intensive outpatient management, or uncontrolled current cognitive status (as confirmed by the specialist; dependence on a caregiver is permitted as long as this is well controlled), severe hepatic comorbidity: liver Child-Pugh grade B-C cirrhosis or acute viral hepatitis, social situations that would limit compliance with study requirements or DIC causing coagulopathy not correctable with factor replacement.
5. Subjects who have had any anti-leukemia treatment prior to entering the study and have not recovered to baseline (except alopecia) or≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and Investigator may be allowed upon agreement with both.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion; anticipated to be 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District

REFERENCES:
- [Derived] Tsai HJ, Hsiao HH, Hsu YT, Liu YC, Kao HW, Liu TC, Cho SF, Feng X, Johnston A, Bomalaski JS, Kuo MC, Chen TY. Phase I study of ADI-PEG20 plus low-dose cytarabine for the treatment of acute myeloid leukemia. Cancer Med. 2021 May;10(9):2946-2955. doi: 10.1002/cam4.3871. Epub 2021 Mar 30. PMID 33787078